CLINICAL TRIAL: NCT00165945
Title: Using 4-D Visualization Software With Magnetic Resonance Images in the Congenital Heart Disease Population
Brief Title: 4-D Visualization Using Magnetic Resonance Imaging (MRI) in the Congenital Heart Disease Population
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, W. James Parks, MD, Assistant Professor, Emory University
Other Study IDs: 075-2004
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Congenital Heart Disease
Keywords: pediatric, cardiology, diagnostic imaging using MRI
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, the investigators wish to use images obtained from standard of care cardiac MRI's performed at Children's Healthcare of Atlanta and transfer the images to a different computer in order to analyze them with a new computer. The investigators are hoping to better their understanding and management of complex congenital heart disease.

DETAILED DESCRIPTION:
All patients enrolled in this study will be receiving standard of care cardiac MRI as prescribed by their physician. These MRI DICOM images will be transferred to a SGI Fuel workstation, where they will be manipulated using the newly developed 4-D Visualization software. No additional scanner time or new imaging sequences are required as presently prescribed sequences and produced data can be analyzed. The workstation is designed to include acceleration hardware for volume rendering, and was developed for advanced cardiac MRI viewing.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a cardiac MRI at Children's Healthcare of Atlanta
* Informed consent
* meet MRI eligibility inclusion criteria

Exclusion Criteria:

* Not having a cardiac MRI
* No informed consent
* not meeting MRI eligibility exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatrics patients in all age groups evaluated with MRI for complex congenital cardiovascular lesions and associated hemodynamics. These are patients coming in for standard of care cardiac MRI's
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2004-06; Primary Completion 2009-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To determine if the 4-D visualization software is beneficial in the investigators' understanding and management of complex congenital heart lesions and their associated hemodynamics/anatomy | throughout study

SECONDARY OUTCOMES:
To study the impact and role of 4-D Visualization on surgical planning and outcome | entire study

CONTACTS AND LOCATIONS:
Overall Officials: W.James Parks, MD, Principal Investigator — Emory University and Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States